CLINICAL TRIAL: NCT04006925
Title: Sodium Oxybate in Treatment-Resistant REM Sleep Behavior Disorder (RBD): A Randomized Placebo-Controlled Trial
Brief Title: Treatment of REM Sleep Behavior Disorder (RBD) With Sodium Oxybate
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 47852
Record Dates: First submitted 2019-06-27; First posted 2019-07-05 (Actual); Results first posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-04

CONDITIONS: REM Sleep Behavior Disorder; Parkinson Disease
Keywords: sodium oxybate
MeSH Terms: conditions — REM Sleep Behavior Disorder; Parkinson Disease | interventions — Sodium Oxybate

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sodium Oxybate (SXB) arm (Active Comparator): Sodium Oxybate (SXB) will be dispensed to the participants.
  Interventions: Drug: Sodium Oxybate
- Placebo (PBO) arm (Placebo Comparator): Placebo will be dispensed to the participants.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Sodium Oxybate — Sodium Oxybate will be titrated up weekly by 1.5g nightly dose increments from an initial 4.5g total nightly dose (which could be given in two unequal doses if needed, or one single dose no greater than 4.5g) to an optimal individual dose based on clinical response on RBD symptoms and tolerance, to a maximum nightly dose of 9g ("flexible dose" period lasting up to 8 weeks). The optimal dose will then be continued for at least 4 weeks ("stable dose").
  Arms: Sodium Oxybate (SXB) arm
Other: Placebo — Placebo will be similar in appearance, smell and flavor to the subjects, so that the investigators and participants will be unable to distinguish it from sodium oxybate.
  Arms: Placebo (PBO) arm

SUMMARY:
This study is the first clinical trial using sodium oxybate for the treatment of REM sleep behavior disorder (RBD). Sodium oxybate is a drug approved by FDA for the treatment of narcolepsy which has been used "off label" to treat patients with severe RBD. This drug has shown to be effective and well tolerated in patients with RBD (Shneerson, 2009; Liebenthal, 2016; Moghadam, 2017).

DETAILED DESCRIPTION:
Rapid eye movement sleep behavior disorder (RBD) is a condition resulting in violent dream-enactment during sleep which affects millions of individuals in the United States, however therapies for RBD are limited and cause significant side effects. As a result, despite using a combination of drugs, a large number of patients with RBD continue to act out violent dreams causing severe self-injuries or injuries to their bed partners. Prior studies and our experience have shown that sodium oxybate can be effective in these cases of treatment-resistant RBD. This study would therefore evaluate the efficacy and tolerance of sodium oxybate in this patient population.

This study is an 8-week trial comparing sodium oxybate versus placebo randomly assigned to patients with treatment-resistant RBD, i.e. individuals who have insufficiently responded or tolerated melatonin and clonazepam. The study uses a double-blind design (participants, staff, and investigators will not know which drug between active drug and placebo is given to participants), and will measure treatment efficacy based on patients, partners and clinicians report, and objective outcomes based on in-home actigraphy and in-lab polysomnography before and after intervention.

ELIGIBILITY:
Inclusion Criteria:

* 40-85 years old
* With or without Parkinson's disease
* Experiencing RBD episodes on average at least 2x/week or 8x/month
* Able to report RBD episodes themselves or via a partner witness

Exclusion Criteria:

* History of falls during ambulation in the last 6 months despite adequate neurologic treatment
* Requirement of an ambulatory device at home
* Inadequately treated symptomatic orthostatic hypotension
* BMI > 35
* Untreated or uncontrolled OSA (4%AHI>15)
* Cognitive impairment resulting in inability to comply with treatment instructions
* Pregnancy

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel During, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shneerson JM. Successful treatment of REM sleep behavior disorder with sodium oxybate. Clin Neuropharmacol. 2009 May-Jun;32(3):158-9. doi: 10.1097/WNF.0b013e318193e394. PMID 19483483
- [Background] Liebenthal J, Valerio J, Ruoff C, Mahowald M. A Case of Rapid Eye Movement Sleep Behavior Disorder in Parkinson Disease Treated With Sodium Oxybate. JAMA Neurol. 2016 Jan;73(1):126-7. doi: 10.1001/jamaneurol.2015.2904. No abstract available. PMID 26595534
- [Background] Moghadam KK, Pizza F, Primavera A, Ferri R, Plazzi G. Sodium oxybate for idiopathic REM sleep behavior disorder: a report on two patients. Sleep Med. 2017 Apr;32:16-21. doi: 10.1016/j.sleep.2016.04.014. Epub 2016 Jun 7. PMID 28366329
- [Derived] During EH, Hernandez B, Miglis MG, Sum-Ping O, Hekmat A, Cahuas A, Ekelmans A, Yoshino F, Mignot E, Kushida CA. Sodium oxybate in treatment-resistant rapid-eye-movement sleep behavior disorder. Sleep. 2023 Aug 14;46(8):zsad103. doi: 10.1093/sleep/zsad103. PMID 37052688

RESULTS

PARTICIPANT FLOW:
Groups:
- Sodium Oxybate (SXB) Arm: For each participant, Sodium Oxybate (SXB) starting at a 4.5g total nightly dose then titrated up weekly by 1.5g increments over 8 weeks to establish their optimal individualized dose (based on their clinical response on RBD symptoms and tolerance). Participant then receive their optimal dose for at least 4 weeks.
- Placebo (PBO) Arm: Placebo similar in appearance, smell and flavor so that it is indistinguishable from sodium oxybate.
Period: Overall Study
Arm/Group | Sodium Oxybate (SXB) Arm | Placebo (PBO) Arm
Started | 12 | 12
Completed | 10 | 12
Not Completed | 2 | 0
Not completed — Side effects | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sodium Oxybate (SXB) Arm | Placebo (PBO) Arm | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.1 (8.2) | 65.4 (7.3) | 65.8 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 9 | 9 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 12 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 12 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 12 | 24
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 24.4 (4.7) | 27.0 (7.6) | 25.7 (6.3)
RBD Symptom Duration [Mean (Standard Deviation); unit: years] | 11.2 (6.9) | 8.4 (4.3) | 9.8 (5.8)
History of Injuries [Count of Participants; unit: Participants] — Injuries related to REM Sleep Behavior Disorder
  Participants | 10 | 12 | 22
Parkinson disease [Count of Participants; unit: Participants] | 6 | 6 | 12
Sleep Apnea [Count of Participants; unit: Participants] | 2 | 5 | 7
Insomnia [Count of Participants; unit: Participants] | 2 | 5 | 7
Current Treatment [Count of Participants; unit: Participants] — Participant's current treatment can include more than 1 medication.
  Participants
    Antidepressant | 4 | 4 | 8
    Clonazepam | 5 | 4 | 9
    Melatonin | 8 | 6 | 14
    Cholinergic | 2 | 1 | 3
    Dopaminergic | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of RBD Episodes in One Month (Per Patient RBD Log)
Description: Patients record any episode of dream enactment, such as talking, shouting, kicking, or punching, etc.
Time Frame: Assessed for 28 days at baseline and during last month of treatment (total treatment period of up to 12 weeks)
Population: Participants with data at each time point are included in the analysis
Measure: Median (Inter-Quartile Range); unit: episodes
Arm/Group | Sodium Oxybate (SXB) Arm | Placebo (PBO) Arm
Number analyzed (Participants) | 12 | 12
episodes
  Baseline | 37.5 [27.5 to 48.5] | 35.0 [28.5 to 45.5]
  Final dose: number analyzed (Participants) | 10 | 12
  Final dose | 23.5 [6.0 to 47.0] | 25.5 [14.5 to 46.0]
Statistical Analysis 1: Comparison: Sodium Oxybate (SXB) Arm; Within group analysis of change from baseline; Test type: Other; p = 0.03, Wilcoxon Signed Rank test — All statistical tests were conducted using a 2-sided alpha level of 0.05; Median Difference (Net) = -23.5, 95% CI 2-sided [-41.0 to -2.0]
Statistical Analysis 2: Comparison: Placebo (PBO) Arm; Within group analysis of change from baseline; Test type: Other; p = 0.11, Wilcoxon Signed Rank test; Median Difference (Net) = -9.0, 95% CI 2-sided [-21.5 to 0.0]
Statistical Analysis 3: Comparison: Sodium Oxybate (SXB) Arm vs Placebo (PBO) Arm; Between group analysis of change from baseline; Test type: Superiority; p = 0.27, Mann Whitney U test — All statistical tests were conducted using a 2-sided alpha level of 0.05; Median Difference (Net) = -14.5, 95% CI 2-sided [-32.0 to 11.3]

2. Primary Outcome: Number of Severe of RBD Episodes in One Month (Per Patient RBD Log)
Description: Patients record any episode of dream enactment, such as talking, shouting, kicking, or punching, etc. Severity is scored from 1 to 3 (1: least severe, 3 most severe):
  1. non injurious behaviors: facial expressions, non-aggressive vocalizations (mumbling, gentle talking, casual conversation, singing, laughing...), twitches, gentle shaking, non-aggressive movements of fingers, arms or legs...;
  2. potentially injurious: punching, kicking, arm flailing or thrashing around, at least one limb or head out of bed, sitting up in bed, crawling, attempting to stand up or leave bed, near falls, cursing, screaming, shouting, yelling, or any behavior requiring bed partner to wake up participant;
  3. injurious: any contact with bed partner (hitting or grabbing), wall or furniture, any fall or leaving bed (doving out, walking, jumping).
  The number of injurious (severe) episodes is reported.
Time Frame: Assessed for 28 days at baseline and during last month of treatment (total treatment period of up to 12 weeks)
Population: Participants with data at each time point are included in the analysis
Measure: Median (Inter-Quartile Range); unit: episodes
Arm/Group | Sodium Oxybate (SXB) Arm | Placebo (PBO) Arm
Number analyzed (Participants) | 12 | 12
episodes
  Baseline | 1.5 [0.5 to 4.0] | 1.5 [0.0 to 3.5]
  Final dose: number analyzed (Participants) | 10 | 12
  Final dose | 0.5 [0.0 to 1.0] | 1.0 [0.0 to 2.5]
Statistical Analysis 1: Comparison: Sodium Oxybate (SXB) Arm; Within group analysis of change from baseline; Test type: Other; p = 0.02, Wilcoxon Signed Rank test — All statistical tests were conducted using a 2-sided alpha level of 0.05; Median Difference (Net) = -1.0, 95% CI 2-sided [-3.0 to 0.0]
Statistical Analysis 2: Comparison: Placebo (PBO) Arm; Within group analysis of change from baseline; Test type: Other; p = 0.83, Wilcoxon Signed Rank test; Median Difference (Net) = 0.0, 95% CI 2-sided [-1.0 to 1.0]
Statistical Analysis 3: Comparison: Sodium Oxybate (SXB) Arm vs Placebo (PBO) Arm; Between group analysis of change from baseline; Test type: Superiority; p = 0.09, Mann Whitney U test — All statistical tests were conducted using a 2-sided alpha level of 0.05; Median Difference (Net) = -1.0, 95% CI 2-sided [-3.5 to 0.0]

3. Secondary Outcome: Number of Responders According to the CGI Efficacy Scale (CGI-E)
Description: Clinical Global Impression-Efficacy index (CGI-E) is a 4x4 rating scale that assesses the therapeutic effect (Marked, Moderate, Minimal, Unchanged or worse) of treatment medication and associated side effects (none, do not significantly interfere with patient's functioning, significantly interfere with patient's functioning, Outweigh therapeutic effect). Therapeutic effect: Marked and Side effects: None is the best. Therapeutic effect: Unchanged or worse and Side effects: outweigh therapeutic effect is the worst. Each combination of an estimated therapeutic effect and side effect is assigned a score from 1-16, 1 being the best, 16 being the worst.
  Participants scoring below 4 were considered to be "responders."
Time Frame: Assessed at week 12 (end of treatment period).
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium Oxybate (SXB) Arm | Placebo (PBO) Arm
Number analyzed (Participants) | 12 | 12
Participants | 10 | 6
Statistical Analysis 1: Comparison: Sodium Oxybate (SXB) Arm vs Placebo (PBO) Arm; Between group analysis of change from baseline; Test type: Superiority; p = 0.08, Mann Whitney U test — All statistical tests were conducted using a 2-sided alpha level of 0.05

4. Secondary Outcome: Number of Responders According to the CGI Improvement Scale (CGI-I)
Description: Clinical Global Impression-Improvement scale (CGI-I) is a 7-point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention and rated as: 1. Very much improved, 2. Much improved, 3. Minimally improved, 4. No change, 5. Minimally worse, 6. Much worse, 7. Very much worse. 1 is the best and 7 is the worst.
  Participants scoring below 4 were considered to be "responders."
Time Frame: Assessed at week 12 (end of treatment period).
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium Oxybate (SXB) Arm | Placebo (PBO) Arm
Number analyzed (Participants) | 12 | 12
Participants | 10 | 7
Statistical Analysis 1: Comparison: Sodium Oxybate (SXB) Arm vs Placebo (PBO) Arm; Between group analysis of change from baseline; Test type: Superiority; p = 0.18, Mann Whitney U test — All statistical tests were conducted using a 2-sided alpha level of 0.05

5. Secondary Outcome: Epworth Sleepiness Scale (ESS) Score
Description: Epworth Sleepiness Scale (ESS) is a scale to assess patients' general level of sleepiness. Patients choose the most appropriate number (0=would never doze, 1=slight chance of dozing, 2=moderate chance of dozing, 3=high chance of dozing) for the each situation: Sitting and reading, Watching TV, Sitting and inactive in a public place, As a passenger in a car for an hour, Lying down to rest in the afternoon, Sitting and talking to someone, Sitting quietly after a lunch, While stopped for a few minutes in the traffic in a car. 0-10: Normal range, 10-12: Borderline, 12-24: Abnormal. Participants recorded their scores for 28 days at baseline and during the 28 days leading up to week 12; scores were then averaged to calculate the score for each time point per participant, and then the median for all participants is reported.
Time Frame: Assessed at baseline and week 12
Population: Participants with data at each time point are included in the analysis
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Sodium Oxybate (SXB) Arm | Placebo (PBO) Arm
Number analyzed (Participants) | 12 | 12
score on a scale
  Baseline | 8.0 [5.5 to 10.0] | 9.5 [4.0 to 10.0]
  Final dose: number analyzed (Participants) | 10 | 12
  Final dose | 5.0 [4.0 to 8.0] | 7.5 [5.0 to 10.5]
Statistical Analysis 1: Comparison: Sodium Oxybate (SXB) Arm; Within group analysis of change from baseline; Test type: Other; p = 0.26, Wilcoxon Signed Rank test — All statistical tests were conducted using a 2-sided alpha level of 0.05; Median Difference (Net) = -1.0, 95% CI 2-sided [-7.0 to 2.0]
Statistical Analysis 2: Comparison: Sodium Oxybate (SXB) Arm vs Placebo (PBO) Arm; Within group analysis of change from baseline; Test type: Other; p = 0.43, Wilcoxon Signed Rank test — All statistical tests were conducted using a 2-sided alpha level of 0.05; Median Difference (Final Values) = -0.5, 95% CI 2-sided [-3.5 to 2.0]
Statistical Analysis 3: Comparison: Sodium Oxybate (SXB) Arm vs Placebo (PBO) Arm; Between group analysis of change from baseline; Test type: Superiority; p = 0.65, Mann Whitney U test — All statistical tests were conducted using a 2-sided alpha level of 0.05; Median Difference (Final Values) = -0.5, 95% CI 2-sided [-4.0 to 3.0]

6. Secondary Outcome: RBD Episode Severity and Frequency During REM Sleep by Quantitative Video-PSG (Polysomnography) Analysis Per 10 Minutes of REM Sleep
Description: The average number of dream-enactment episodes (resulting in motor behaviors, or movements) weighted for severity. Frequency and severity were calculated as the sum of RBD episodes (frequency) times severity (mild = 1; moderate = 5, severe = 10) occurring over one night's sleep, then averaged to calculate the number of episodes per 10 minutes of REM sleep.
Time Frame: Assessed at baseline and week 12 (average approximately 8 hours to assess at each time point)
Population: Participants with data available at the respective time points are presented.
Measure: Mean (Standard Deviation); unit: episodes*severity per 10 minutes of REM
Arm/Group | Sodium Oxybate (SXB) Arm | Placebo (PBO) Arm
Number analyzed (Participants) | 8 | 10
episodes*severity per 10 minutes of REM
  Baseline | 13.2 (12.3) | 10.1 (8.4)
  Final dose: number analyzed (Participants) | 7 | 9
  Final dose | 7.2 (7.4) | 10.5 (10.0)
Statistical Analysis 1: Comparison: Sodium Oxybate (SXB) Arm; Within group analysis of change from baseline; Test type: Other; p = 0.23, Unpaired T-test — All statistical tests were conducted using a 2-sided alpha level of 0.05; Mean Difference (Net) = -6.2, 95% CI 2-sided [-15.2 to 1.7]
Statistical Analysis 2: Comparison: Placebo (PBO) Arm; Within group analysis of change from baseline; Test type: Other; p = 0.95, Unpaired T-test — All statistical tests were conducted using a 2-sided alpha level of 0.05; Mean Difference (Net) = 0.2, 95% CI 2-sided [-4.6 to 4.5]
Statistical Analysis 3: Comparison: Sodium Oxybate (SXB) Arm vs Placebo (PBO) Arm; Between group analysis of change from baseline; Test type: Superiority; p = 0.22, Paired T-test — All statistical tests were conducted using a 2-sided alpha level of 0.05; Mean Difference (Net) = -6.4, 95% CI 2-sided [-16.2 to 3.1]

7. Secondary Outcome: Change in Ambulatory Measures of Movements During Sleep Using Actigraphy
Description: Measure of "activity score" using in-home 4-week actigraphy
Time Frame: Assessed for 28 days at baseline and during last month of treatment (total treatment period of up to 12 weeks)
Population: Analysis was not possible because the data that were collected were corrupted and uninterpretable.
Arm/Group | Sodium Oxybate (SXB) Arm | Placebo (PBO) Arm
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 12 weeks
Arm/Group | Sodium Oxybate (SXB) Arm | Placebo (PBO) Arm
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 5/12 | 0/12
Other Adverse Events (participants affected / at risk) | 7/12 | 2/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sodium Oxybate (SXB) Arm (N=12) | Placebo (PBO) Arm (N=12)
Myoclonus episode (Musculoskeletal and connective tissue disorders) | 1 | 0
Sleep terror (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sodium Oxybate (SXB) Arm (N=12) | Placebo (PBO) Arm (N=12)
Anxiety (Psychiatric disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Auditory hallucination (Psychiatric disorders) | 1 | 0
Brain fog (General disorders) | 2 | 0
Enuresis (Renal and urinary disorders) | 1 | 0
Gastrointestinal discomfort (Gastrointestinal disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Hot flashes (General disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Sensation of being "wired" (General disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Anorexia (Psychiatric disorders) | 2 | 0
Catathrenia (General disorders) | 1 | 0
Increased sweating (General disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Dysgeusia (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-07-08): https://cdn.clinicaltrials.gov/large-docs/25/NCT04006925/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-11): https://cdn.clinicaltrials.gov/large-docs/25/NCT04006925/SAP_001.pdf